CLINICAL TRIAL: NCT02671214
Title: The Effect of Selected Fibres and Flours in Flat Bread on Post-prandial Blood Glucose Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 10020V
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: guar gum; konjac mannan; blood glucose; legume flour
MeSH Terms: interventions — Bc-4 active principle; pTAC5 protein, Arabidopsis; pTAC10 protein, Arabidopsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Control (Placebo Comparator): 100 g high fibre flour
  Interventions: Other: Control
- Active 1 (Active Comparator): 85 g high fibre flour + 15 g legume flour
  Interventions: Other: Active 1
- Active 2 (Active Comparator): 98 g high fibre flour + 2 g guar gum
  Interventions: Other: Active 2
- Active 3 (Active Comparator): 88 g high fibre flour + 2 g guar gum + 10 g legume flour
  Interventions: Other: Active 3
- Active 4 (Active Comparator): 83 g high fibre flour + 2 g guar gum + 15 g legume flour
  Interventions: Other: Active 4
- Active 5 (Active Comparator): 96 g high fibre flour + 4 g guar gum
  Interventions: Other: Active 5
- Active 6 (Active Comparator): 86 g high fibre flour + 4 g guar gum + 10 g legume flour
  Interventions: Other: Active 6
- Active 7 (Active Comparator): 81 g high fibre flour + 4 g guar gum + 15 g legume flour
  Interventions: Other: Active 7
- Active 8 (Active Comparator): 94 g high fibre flour + 6 g guar gum
  Interventions: Other: Active 8
- Active 9 (Active Comparator): 98 g high fibre flour + 2 g konjac mannan
  Interventions: Other: Active 9
- Active 10 (Active Comparator): 96 g high fibre flour + 4 g konjac mannan
  Interventions: Other: Active 10
- Active 11 (Active Comparator): 100 g low fibre flour
  Interventions: Other: Active 11

INTERVENTIONS:
Other: Control — 100 g high fibre flour
  Arms: Control
Other: Active 2 — 98 g high fibre flour + 2 g guar gum
  Arms: Active 2
Other: Active 3 — 88 g high fibre flour + 2 g guar gum + 10 g legume flour
  Arms: Active 3
Other: Active 4 — 83 g high fibre flour + 2 g guar gum + 15 g legume flour
  Arms: Active 4
Other: Active 5 — 96 g high fibre flour + 4 g guar gum
  Arms: Active 5
Other: Active 6 — 86 g high fibre flour + 4 g guar gum + 10 g legume flour
  Arms: Active 6
Other: Active 7 — 81 g high fibre flour + 4 g guar gum + 15 g legume flour
  Arms: Active 7
Other: Active 8 — 94 g high fibre flour + 6 g guar gum
  Arms: Active 8
Other: Active 9 — 98 g high fibre flour + 2 g konjac mannan
  Arms: Active 9
Other: Active 10 — 96 g high fibre flour + 4 g konjac mannan
  Arms: Active 10
Other: Active 11 — 100 g low fibre flour
  Arms: Active 11
Other: Active 1 — 85 g high fibre flour + 15 g legume flour
  Arms: Active 1

SUMMARY:
Identify one or more flat bread mixes that produce a reduction in positive incremental area under the curve (iAUC) of post-prandial glucose relative to the control product.

DETAILED DESCRIPTION:
This study was a double-blind, randomised, balanced incomplete block design exploratory study of efficacy, with 11 active treatments compared to a control product in 42 healthy subjects to see if a mix of active ingredients (viscous fibres and flours) lowered the post-prandial glucose (PPG) response in capillary blood (finger prick) over a two and three hours period, relative to the control product. Every subject received the control and 4 out of the 11 treatments on five separate test days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 20 and ≤ 25.0 kg/m2.
* Apparently healthy: no medical conditions which might affect study measurements (as judged by the study physician).
* A fasting blood glucose value between 3.5 - 5.6 mmol/litre at screening (measured by finger prick).

Exclusion Criteria:

* Use of medication which interferes with study measurements (as judged by the study physician).
* Reported dietary habits: medically prescribed diet, slimming diet, not used to eat 3 meals a day, vegetarian.
* Reported weight loss/gain (>10%) in the last six month before the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Positive incremental area under the curve (iAUC) | 120 minutes

SECONDARY OUTCOMES:
Positive incremental area under the curve (iAUC) | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hull, Principal Investigator — Leatherhead Food Research UK
Locations (1):
- Leatherhead Food Research UK, Leatherhead, Randalls Road, Surrey, United Kingdom

REFERENCES:
- [Derived] Boers HM, MacAulay K, Murray P, Seijen Ten Hoorn J, Hoogenraad AR, Peters HPF, Vente-Spreeuwenberg MAM, Mela DJ. Efficacy of different fibres and flour mixes in South-Asian flatbreads for reducing post-prandial glucose responses in healthy adults. Eur J Nutr. 2017 Sep;56(6):2049-2060. doi: 10.1007/s00394-016-1242-9. Epub 2016 Jun 21. PMID 27324141